CLINICAL TRIAL: NCT00987753
Title: A PhaseI/II Study Evaluating the Safety, Tolerability, and Maximally Tolerated Dose of L-377202 Administered Once Every 3 Weeks
Brief Title: Study Evaluating the Safety and Tolerability of L-377202
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Michael James Bertram, Proffessor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F990224004; UAB 9902; NCT00004185 (obsolete NCT alias)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hormone Refractory Prostate Cancer; Prostate Cancer
Keywords: L-377202, prostate cancer, PSA
MeSH Terms: conditions — Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- infusion of L-377202 (Experimental)
  Interventions: Drug: L-377202

INTERVENTIONS:
Drug: L-377202 — For each cycle, L-377202 will be administered as a 30-minute infusion every 3 weeks. The starting dose will be 20 mg/m2/week. Doses will be doubled until a patient experiences a greater than or equal to Grade 2 toxicity.

SUMMARY:
The primary purpose of this study is to (1) determine the maximally tolerated dose (MTD) of L-377202 administered once every 3 weeks, (2) evaluate the safety and tolerability of L-377202 including the dose-limiting adverse effects of treatment with L-377202, and (3) assess the pharmacokinetics of various doses of L-377202 and the plasma profile of liberated doxorubicin and leu-doxorubicin.

DETAILED DESCRIPTION:
This is an open, nonrandomized, rising-dose study in patients with hormone refractory prostate cancer. Patients will be treated with L-377202 once every three weeks. Plasma concentrations of L-377202, liberated doxorubicin, and leu-doxorubicin will be obtained at defined time intervals throughout the study. At least 1 patient will be treated at each dose level until there is evidence of greater than or equal to Grade 2 drug-related toxicity. Each patient will be treated at only 1 dose level, although multiple cycles may be administered until signs of disease progression or unacceptable toxicity are evident. Doses will be doubled for each subsequent cohort of patients until evidence of greater than or equal to Grade 2 drug-related toxicity. Upon documentation of greater than or equal to Grade 2 drug-related toxicity, subsequent dose escalations will proceed along the modified Fibonacci scale and enroll at least 3 patients per dose level until 1 patient experiences dose-limiting toxicity (DLT).

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least an 18-year-old male and has histologically documented, progressive carcinoma of the prostate which is refractory to hormonal manipulation. Progressive disease may be documented by new lesions on bone scan, increase in radiologically measurable disease, or an increase in PSA (at least 50% increase from nadir confirmed twice and measured at least 2 weeks apart.)
* An appropriate interval of time has passed since alteration of any hormonal therapy (e.g., 4 weeks for steroids, LHRH agonists, flutamide or megestrol acetate and 6 weeks for nilutamide and bicalutamide).
* Patient has a serum PSA of 20 ng/mL or higher.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Patients has a life expectancy of >3 months.
* Patient understands and agrees to participate in the study by providing written informed consent.

Exclusion Criteria:

* Patient is mentally or legally incapacitated at the time of the study or has a history (less than 5 years prior to entry) of drug or alcohol abuse or is currently a user (including "recreational use") of any illicit drugs.
* Patient has known HIV or a known HIV-related malignancy.
* Patient has participated in another study (including FDA approved drugs for a non-FDA approved indication) of an investigational agent within the last 4 weeks.
* Patient requires treatment or is anticipated to require treatment with Cyclosporine, Phenobarbital, phenytoin, or streptozocin.
* Patient has received tumor directed immunologic therapy, radiation therapy, surgery, or chemotherapy within 4 weeks of the study. However, patients who are receiving thyroid replacement therapy may be included. For mitomycin or nitrosourea, there must be a 6-week treatment free interval.
* Patient has received strontium treatment within 12 weeks prior to treatment.
* Patient is anticipated to require immunologic therapy, radiation therapy, surgery, or chemotherapy during the study.
* Patient has received high-dose chemotherapy with stem cell rescue.
* Patient has a history of significant cardiac dysrhythmias (Grade 3 or higher excluding atrial fibrillation).
* Patient has recently had (within 6 months) a myocardial infarction, unstable angina, or congestive heart failure.
* Patient has an abnormal PT (INR) or a PTT (>1.2 times normal). Low-dose warfarin (1 to 2 mg P.O. q.d.) or heparin (the equivalent of 5000 IU SQ b.i.d.) administered to maintain catheter patency is acceptable. Patients administered higher doses of anticoagulants may be considered on an individual basis pending discussion between the clinical monitor and investigator. Such patients will require more intensive monitoring of PT (INR) and aPTT (at least every other day).
* Patient has an absolute neutrophil count <1500/mm3 or platelet count <100,000/mm3 or hemoglobin <9 gm/dL, bilirubin >1.5 times normal or ALT or AST >2.5 times normal or creatinine >1.5 times normal.
* Patient has an active infection.
* Patient has an active (edema, progressive disease, or clinical neurologic symptoms) metastatic CNS lesion.
* Patient has received the equivalent of >180 mg/m2 of doxorubicin or >40 mg/m2 mitoxantrone.
* Patient has left ventricular ejection fraction (LVEF) <45%.
* Patient has received radiation to >25% of his total bone marrow.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1999-03; Primary Completion 2000-09 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the administration of L-377202 every three weeks in patients with hormone refractory prostate cancer | Every 3 weeks until disease progression or unacceptable toxicity

SECONDARY OUTCOMES:
Evaluation of the radiologic and/or PSA responses to L-377202 treatment | Every 3 weeks until disease progression or unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: John Rinehart, M.D., Principal Investigator — University of Alabama at Birmingham (no longer employee); Scot Ebbinghaus, M.D., Principal Investigator — University of Alabama at Birmingham (no longer employee)
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States